CLINICAL TRIAL: NCT02438163
Title: Study of Neuroplasticity on Depressed Patients Versus Healthy Subjects : Modulation of the MEP Size Induced by Theta Burst Stimulation
Brief Title: Study of Neuroplasticity on Depressed Patients : Modulation of MEP Induced by Theta Burst Stimulation
Acronym: DEPLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Principal Investigator, VIGNAUD Philippe, medical doctor, Hôpital le Vinatier
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HopitalVinatier
Record Dates: First submitted 2015-04-08; First posted 2015-05-08 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Depression
Keywords: Theta Burst Stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with MDD (Experimental): the group of depressed patients undergo 2 Theta Burst Stimulations : iTBS and cTBS. There is one session per stimulation. Cerebral Plasticity is measured after each stimulation for each session
  Interventions: Device: Theta Burst Stimulation
- healthy Controls (Experimental): the group of healthy controls undergo 2 Theta Burst Stimulations : iTBS and cTBS. There is one session per stimulation. Cerebral Plasticity is measured after each stimulation for each session
  Interventions: Device: Theta Burst Stimulation

INTERVENTIONS:
Device: Theta Burst Stimulation — During the first session, After determining the parameters of stimulation (stimulated target : part of the left motor cortex responsible for the contraction of the right first dorsal interosseous muscle ; Activity Motor Threshold (AMT) ; Intensity of Stimulation providing a Motor Evoked Potential (MEP) with an Amplitude of 1mV (MEP 1mV)), a Baseline consisting of 15 MEP (intensity MEP 1mV) is measured. Then each subjet receive a TBS protocol (cTBS or iTBS) (intensity of stimulation 80% of AMT). After receiving the stimulation, sets containing 10 MEP are regularly measured by each subject.
  During a second session, the same protocol is done again with the other TBS stimulation (cTBS or iTBS) the subject didn't get during the first session.

SUMMARY:
Neuroplasticity is supposed to be altered in patients suffering from a Major Depressive Disorder (MDD). Transcranial Magnetic Stimulation is a medical device which measures cerebral plasticity. Several parameters of cortical excitability are available for that purpose. These parameters are altered on patients wth MDD and these modifications are corrected after treatment. Therefore results in the studies are very heterogeneous. Theta Burst Stimulation (TBS) is a type a Transcranial Magnetic Stimulation (TMS) protocol and can induce cerebral plasticity. The cerebral plasticity induced by TBS was measured on a group of patients suffering from Asperger's disease (ASD) versus a control group. The plasticity was significantly different in patients with ASD. The aim of our study is to study the neuroplasticity induced by TBS on a patients with MDD.

DETAILED DESCRIPTION:
The study is lead with patients suffering from a MDD. All patients are drug free. Patients are compared to a control group of healthy subjects The protocol has 2 sessions. During the first session, After determining the parameters of stimulation (stimulated target : part of the left motor cortex responsible for the contraction of the right first dorsal interosseous muscle ; Activity Motor Threshold (AMT) ; Intensity of Stimulation providing a Motor Evoked Potential (MEP) with an Amplitude of 1mV (MEP 1mV)), a Baseline consisting of 15 MEP (intensity MEP 1mV) is measured. Then each subjet receive a TBS protocol (cTBS or iTBS) (intensity of stimulation 80% of AMT). After receiving the stimulation, sets containing 10 MEP are regularly measured by each subject.

During a second session, the same protocol is done again with the other TBS stimulation (cTBS or iTBS) the subject didn't get during the first session.

A neuronavigation device is used to determine precisely the area of stimulation.

ELIGIBILITY:
Inclusion Criteria:

Subjects with MDD

* MDD according to definition provided by the DSM V
* No antidepressant Healthy Controls
* No present psychiatric disease

Exclusion Criteria:

* depression with Melancholic features
* pregnancy
* contra indication in the use of TMS (personal history of epilepsy, deep brain stimulation, vague nerve stimulation, pace maker, intracerebral lesion, pieces of metal Inside of the brain)
* diseases with neurological effects (multiple sclerosis, Parkinson disease, HIV...)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03-21 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Time needed for MEP amplitude to return to Baseline after TBS | Baseline, up to 120 minutes post TBS
  The primary outcome is determined by measuring the MEP size at 5/10/20/30/40/50/60/75/90/105/120 min post TBS. Then we determine when the MEP size comes back to the Baseline measure

SECONDARY OUTCOMES:
Size-effect of modification of MEP size after TBS | The secondary outcome is determined by measuring the MEP size 5/10/20/30/40/50/60/75/90/105/120 min post TBS

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel POULET, MD PhD, Study Director — Hôpital le Vinatier
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vignaud P, Damasceno C, Poulet E, Brunelin J. Impaired Modulation of Corticospinal Excitability in Drug-Free Patients With Major Depressive Disorder: A Theta-Burst Stimulation Study. Front Hum Neurosci. 2019 Feb 26;13:72. doi: 10.3389/fnhum.2019.00072. eCollection 2019. PMID 30863297